# National Longitudinal Cohort of Hematological Diseases - Blood Disease Infection (NICHE- BDI)

Applicant: Institute of Hematology & Blood Diseases Hospital

Version: 1.0

Date: 7-Dec-2022

National Longitudinal Cohort of Hematological Diseases- Blood Disease Infection (NICHE- BDI)

### Background

Hematological diseases are disorders of the blood and hematopoietic organs. The current hematological cohorts are mostly based on single-center or multi-center cases, or cohorts with limited sample size in China. There is a lack of comprehensive and large-scale prospective cohort studies in hematology.

### Objectives

The objectives of this study are to investigate the incidence and risk factors of blood disease infection and to analyze the treatment methods, prognosis and medical expenses of these patients in China.

## Subjects

Patients who were diagnosed with blood disease infection in the investigating hospitals from December 7, 2022.

### Method

The NICHE-BDI will collect basic information, diagnostic and treatment information, as well as medical expense information of patients from medical records. The study will use questionnaire to measure the exposure of patients, and prospectively follow-up to collect the prognosis information.

# **Statistical Analysis Plan**

Statistical analyses will be performed using SAS 9.4 (SAS Institute Inc., Cary, NC, USA) software. For the categorical variables, the results will be presented as counts and percentages. The differences between groups were compared with Chi-square test or Fisher's exact test. For continuous variables, mean  $\pm$  SD or median (P25, P75) will be presented according to the distributions. The differences between groups were compared with ANOVA or Wilcoxon rank-sum test. For time-to-event variables, the incidences of events were described using the Kaplan-Meier method and compared between groups using the log-rank test. Cox proportional hazard regression modes were used for multivariate analyses. A P-value of less than 0.05 was considered to indicate statistical significance.